CLINICAL TRIAL: NCT04682587
Title: A Panel-Based Chart Review Study to Examine the Effects of Axitinib Dose Reduction and Interruption for Adverse Event Management Among Patients Receiving First-Line Axitinib in Combination With Immune-Oncology Drugs for the Treatment of Advanced Renal Cell Carcinoma
Brief Title: To Examine the Effects of Axitinib Dose Reduction and Interruption for Adverse Event Management Among Patients Receiving Axitinib in for the Treatment of Advanced Renal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A4061097
Record Dates: First submitted 2020-12-10; First posted 2020-12-24 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Renal Cell Carcinoma
Keywords: Advanced Renal Cell Carcinoma (aRCC)
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Axitinib; avelumab; pembrolizumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Axitinib — Inlyta, axitinib
Drug: Avelumab — Avelumab, Bavencio
Drug: Pembrolizumab — Pembrolizumab, Keytruda

SUMMARY:
To assess how dose reductions or treatment interruptions related to axitinib can be implemented to manage and resolve adverse events occurring among patients with advanced renal cell carcinoma treated with first-line axitinib in combination with avelumab or pembrolizumab

DETAILED DESCRIPTION:
The specific objectives of the study are as follows:

Describe incident adverse events (AEs) experienced among patients with advanced RCC who received first-line axitinib in combination with immuno-oncology (IO) therapies.

* Type and seriousness of AEs (ie, diarrhea, fatigue, hypertension, nausea, palmar plantar erythrodysesthesia [hand-foot syndrome]).
* Proportion of patients who experienced repeated AEs.
* Time from treatment initiation to AE onset, overall and by type and seriousness of AEs.

Among patients with advanced RCC who developed incident AEs while receiving first line axitinib in combination with IO therapies, characterize and describe management strategies for AEs, stratified by type and seriousness of AEs.

* Proportion of patients who used each of the following management strategies:
* No action for axitinib and IO therapy;
* No action for axitinib, but treatment modification for IO therapy (ie, treatment interruption, treatment discontinuation);
* Axitinib dose reduction, but no action for IO therapy;
* Axitinib treatment interruption, but no action for IO therapy;
* Axitinib treatment discontinuation, but no action for IO therapy;
* Axitinib dose reduction, and treatment modification for IO therapy;
* Axitinib treatment interruption, and treatment modification for IO therapy;
* Axitinib treatment discontinuation, and treatment modification for IO therapy.
* Average axitinib dose reduction (absolute and percentage change), where applicable.
* Duration of treatment interruption, where applicable.

Assess the frequency of and time to AE resolution (from AE onset and initiation of management strategy, separately) among patients with advanced RCC who developed incident AEs while receiving first-line axitinib in combination with IO therapies according to different management strategies implemented, stratified further by type and seriousness of AEs, as allowed by sample size.

The above objectives will also be conducted for repeated AEs of the same type

ELIGIBILITY:
Inclusion Criteria:

Physicians meeting the following criteria will be invited to participate in the chart review study:

* Specialty in oncology
* Access to complete medical records for at least one patient with advanced RCC who meets the patient eligibility criteria

Eligible oncologists will be asked to select up to three patients meeting the following criteria for inclusion in the chart review study:

* Confirmed diagnosis with advanced RCC
* Treated with first-line axitinib/IO combination therapy at or after diagnosis
* Experienced at least one AE (i.e., diarrhea, fatigue, nausea, hypertension, and palmar-plantar erythrodysesthesia [hand-foot syndrome]) while treated with axitinib/IO combination therapy
* Age 18 years or older at the time of advanced RCC diagnosis
* Initiated axitinib/IO combination therapy at least 3 months prior to the start date of medical chart abstraction to ensure sufficient follow-up time

Exclusion Criteria:

There are no exclusion criteria for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with aRCC
Sampling Method: Non-Probability Sample
Enrollment: 481 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Zakharia Y, Huynh L, Du S, Chang R, Pi S, Sundaresan S, Duh MS, Zanotti G, Thomaidou D. Impact of Therapy Management on Axitinib-Related Adverse Events in Patients With Advanced Renal Cell Carcinoma Receiving First-Line Axitinib + Checkpoint Inhibitor. Clin Genitourin Cancer. 2023 Oct;21(5):e343-e351. doi: 10.1016/j.clgc.2023.03.017. Epub 2023 Apr 3. PMID 37087399
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A4061097

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of participants with advanced Renal cell carcinoma (RCC) who received first line therapy of Axitinib in combination with Immuno-oncology (IO) therapy was observed in this study. Oncologists abstracted data from medical charts of eligible participants using an online electronic case report form (eCRF). Abstracted data was evaluated over 1.5 months of this retrospective study.
Groups:
- Axitinib + IOs: Participants with advanced RCC who received first-line axitinib in combination with IO (avelumab or pembrolizumab) in real world per routine clinical practice, their data were abstracted from medical charts and observed during this retrospective study.
Period: Overall Study
Arm/Group | Axitinib + IOs
Started | 481
Completed | 481
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All eligible participants whose data were extracted from medical records and observed in the study.
Arm/Group | Axitinib + IOs
Number analyzed (Participants) | 481
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161
  Male | 320
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 76
  White | 358
  Unknown or Not Reported | 6
  Missing | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Different Type of Adverse Events
Description: An AE was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship to it.Index date was defined as the initiation of first-line axitinib (used in combination with IO therapy) on or after May 2019, which marked FDA approval of axitinib in combination with avelumab for first-line advanced RCC treatment. Observation period was time from index date to the earliest of initiation of a second line therapy, death, loss to follow-up, or date of chart abstraction. Data, index date, and observation period were on the basis of data extracted from medical charts of participants.
Time Frame: Observation period of maximum up to 7.1 months; duration of this retrospective study was approximately 1.5 months
Population: All eligible participants whose data were extracted from medical records and observed in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib + IOs
Number analyzed (Participants) | 481
Participants
  Fatigue | 232
  Diarrhea | 184
  Nausea | 141
  Hypertension | 106
  Palmar-plantar erythrodysesthesia | 54

2. Primary Outcome: Number of Participants With Serious Adverse Events
Description: AE was considered serious when it: resulted in death, life-threatening, requires in-participant hospitalization or prolongation of existing hospitalization, resulted in a persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event that may jeopardize the participant or may require intervention to prevent one of the outcomes listed above. Index date was defined as the initiation of first-line axitinib (used in combination with IO therapy) on or after May 2019, which marked FDA approval of axitinib in combination with avelumab for first-line advanced RCC treatment. Observation period was time from index date to the earliest of initiation of a second line therapy, death, loss to follow-up, or date of chart abstraction. Data, index date, and observation period were on the basis of data extracted from medical charts of participants.
Time Frame: 6 months
Population: All eligible participants whose data were extracted from medical records and observed in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib + IOs
Number analyzed (Participants) | 481
Participants | 130

3. Primary Outcome: Duration From Treatment Initiation to Onset of Adverse Events
Description: An AE was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship to it. In this outcome measure time from index date to occurrence of incidence of any AE is reported. Index date was defined as the initiation of first-line axitinib (used in combination with IO therapy) on or after May 2019, which marked FDA approval of axitinib in combination with avelumab for first-line advanced RCC treatment. Observation period was time from index date to the earliest of initiation of a second line therapy, death, loss to follow-up, or date of chart abstraction. Data, index date, and observation period were on the basis of data extracted from medical charts of participants.
Time Frame: Observation period of maximum up to 7.1 months; duration of this retrospective study was approximately 1.5 months
Population: All eligible participants whose data were extracted from medical records and observed in the study.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Axitinib + IOs
Number analyzed (Participants) | 481
Months | 1.0 [0.3 to 2.0]

4. Primary Outcome: Duration of Adverse Events From Onset to Resolution
Description: The time to resolution from AE onset and from initiation of management strategy was calculated for all AEs experienced including repeated AEs. The time to resolution of AE (from the onset of AE and from the initiation of management strategies) was separately estimated using Kaplan-Meier analysis; median time to event will be reported. Index date was defined as the initiation of first-line axitinib (used in combination with IO therapy) on or after May 2019, which marked FDA approval of axitinib in combination with avelumab for first-line advanced RCC treatment. Observation period was time from index date to the earliest of initiation of a second line therapy, death, loss to follow-up, or date of chart abstraction. Data, index date, and observation period were on the basis of data extracted from medical charts of participants.
Time Frame: Observation period of maximum up to 7.1 months; duration of this retrospective study was approximately 1.5 months
Population: All eligible participants whose data were extracted from medical records and observed in the study.
Measure: Median (Inter-Quartile Range); unit: Days
Units Other Than Participants: Adverse Events
Arm/Group | Axitinib + IOs
Number analyzed (Participants) | 481
Number analyzed (Adverse Events) | 729
Days
  Overall | 21.0 [9.0 to 33.0]
  Severe AE's: number analyzed (Adverse Events) | 102
  Severe AE's | 17.0 [6.0 to 31.0]

5. Primary Outcome: Number of Adverse Events Classified According to Type of Management Strategy
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with the study treatment. Index date was defined as the initiation of first-line axitinib (used in combination with IO therapy) on or after May 2019, which marked FDA approval of axitinib in combination with avelumab for first-line advanced RCC treatment. Observation period was time from index date to the earliest of initiation of a second line therapy, death, loss to follow-up, or date of chart abstraction. Data, index date, and observation period were on the basis of data extracted from medical charts of participants.
Time Frame: Observation period of maximum up to 7.1 months; duration of this retrospective study was approximately 1.5 months
Population: All eligible participants whose data were extracted from medical records and observed in the study.
Measure: Number; unit: Adverse Events
Units Other Than Participants: Adverse Events
Arm/Group | Axitinib + IOs
Number analyzed (Participants) | 481
Number analyzed (Adverse Events) | 729
Adverse Events
  No Action | 198
  Axitinib modifications (with or without supportive care) | 251
  Axitinib modifications with IO treatment modification: number analyzed (Adverse Events) | 251
  Axitinib modifications with IO treatment modification | 96

6. Primary Outcome: Duration of Treatment Interruption for Axitinib
Description: Duration of treatment interruption was calculated as the total days of treatment interruption. Index date was defined as the initiation of first-line axitinib (used in combination with IO therapy) on or after May 2019, which marked FDA approval of axitinib in combination with avelumab for first-line advanced RCC treatment. Observation period was time from index date to the earliest of initiation of a second line therapy, death, loss to follow-up, or date of chart abstraction. Data, index date, and observation period were on the basis of data extracted from medical charts of participants.
Time Frame: Observation period of maximum up to 7.1 months; duration of this retrospective study was approximately 1.5 month
Population: All eligible participants whose data were extracted from medical records and observed in the study.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Axitinib + IOs
Number analyzed (Participants) | 481
Days | 13.0 [7.0 to 21.0]

7. Primary Outcome: Maximum Axitinib Dose Reduction
Description: Maximum axitinib dose reduction was calculated as the difference between axitinib dose at AE onset and the minimum axitinib dose recorded between the date of AE onset and either the date of AE resolution (if the AE had a reported resolution date) or the end of follow up (if the AE did not have a reported resolution date).Index date was defined as the initiation of first-line axitinib (used in combination with IO therapy) on or after May 2019, which marked FDA approval of axitinib in combination with avelumab for first-line advanced RCC treatment. Observation period was time from index date to the earliest of initiation of a second line therapy, death, loss to follow-up, or date of chart abstraction. Data, index date, and observation period were on the basis of data extracted from medical charts of participants.
Time Frame: Observation period of maximum up to 7.1 months; duration of this retrospective study was approximately 1.5 months
Population: All eligible participants whose data were extracted from medical records and observed in the study.
Measure: Median (Inter-Quartile Range); unit: Milligrams twice daily
Arm/Group | Axitinib + IOs
Number analyzed (Participants) | 481
Milligrams twice daily | 3.0 [2.0 to 3.5]

ADVERSE EVENTS:
Time Frame: Observation period of maximum up to 7.1 months; duration of this retrospective study was approximately 1.5 months
Description: An AE term may be reported as both a serious and non-serious AE but are distinct events. An AE may be serious for 1 participant and non-serious for another participant, or a participant may have experienced both a serious and non-serious episode of the same event. AEs were reported as per participant's medical records. There was no specific medical dictionary.
Arm/Group | Axitinib + IOs
All-Cause Mortality (participants affected / at risk) | 32/481
Serious Adverse Events (participants affected / at risk) | 130/481
Other Adverse Events (participants affected / at risk) | 265/481
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + IOs (N=481)
Fatigue (General disorders) | 21
Diarrhoea (Gastrointestinal disorders) | 51
Nausea (Gastrointestinal disorders) | 17
Hypertension (Vascular disorders) | 28
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 13
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + IOs (N=481)
Fatigue (General disorders) | 107
Diarrhoea (Gastrointestinal disorders) | 55
Nausea (Gastrointestinal disorders) | 49
Hypertension (Vascular disorders) | 41
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/87/NCT04682587/Prot_SAP_000.pdf